CLINICAL TRIAL: NCT01995812
Title: Ola Hou i ka Hula: A Pilot Study to Investigate Hula and Hypertension Control
Brief Title: Ola Hou i ka Hula: Hula and Hypertension
Acronym: Ola Hou
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Principal Investigator, Joseph Keawe'aimoku Kaholokula, Chair and Associate Professor, University of Hawaii
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ola Hou i ka Hula
Record Dates: First submitted 2013-11-18; First posted 2013-11-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

ARMS (2):
- Hula and heart health education (Experimental): 12 weeks of hula classes, 2 times a week for one hour. An additional 3 hours of heart health education was given to participants
  Interventions: Behavioral: Hula and heart health education
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Hula and heart health education
  Arms: Hula and heart health education

SUMMARY:
Physical activity is an important lifestyle modification for individuals with high blood pressure. It is part of national cardiac care guidelines for hypertension management that recommends, along with prescribing medication, lifestyle modification be promoted for improved dietary intake, and participation in about 150 minutes of moderate exercise a week. Native Hawaiians and other Pacific peoples (NHPP) have among the highest risk for the heart disease, with mortality rates twice other ethnic groups. In many minority populations, including NHPP, hypertension develops at an early age, is more severe and is less likely to be controlled. Despite the ability of physical activity to reduce blood pressure, the majority of U.S. population, do not meet physical activity recommendations and new interventions that can improve accessibility and adherence, particularly among at-risk minority populations are needed.

In this research, Hypertension and Hula: Ola Hou Pilot Study, we plan to evaluate a culturally relevant intervention that uses hula and is consistent with the goals of recommended physical activity for improved lifestyle - moderate-intensity, prolonged physical activity cumulatively at about 150 minutes per week. Hula, the traditional dance form of Native Hawaiians, is commonly practiced in Hawai'i as a cultural practice, form of creative expression, and exercise that is structured on controlled, rhythmic movements. Combining aspects of meditation, music, self-awareness with low-impact aerobic exercise, traditional hula may be particularly suitable to individuals with limited mobility and fitness and within the recommended paradigm for exercise training and secondary prevention of coronary artery disease (CAD). We anticipate a hula and heart health education program will be particularly appealing to Native Hawaiians and other Pacific people (NHPP) including Pacific Islanders and Filipino who suffer from a significant disparity in cardiovascular health.

Specifically, we will determine if individuals with poorly managed hypertension and randomized to a 12-week hula and heart health education intervention will demonstrate better blood pressure levels, functional capacity, and exercise tolerance (6-minute walk test) than individuals randomized to a usual care group. We will also assess if the individuals in the hula intervention report better health-related quality of life, stress management, perceptions of discrimination, and exercise self efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age > 18) with blood pressure >140/90 or >130/80 if also diagnosed with diabetes
* Under a physicians care for hypertension for at least 6 months
* Prescribed 2-3 hypertension medications
* Independently ambulatory
* Approval of participation from primary care physician or cardiologist

Exclusion Criteria:

* Prescribed more than 4, or only 1 hypertension medication
* Severe cognitive dysfunction precluding informed consent and understanding of hula
* Pregnancy at time or during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Reduction of systolic blood pressure in hypertensive participants | 3 months

SECONDARY OUTCOMES:
Health-related quality of life | 3 months
  Additional surveys given to participants to measure psychosocial factors.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hawaii, John A Burns School of Medicine, Department of Native Hawaiian Health, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Kaholokula JK, Look M, Mabellos T, Zhang G, de Silva M, Yoshimura S, Solatorio C, Wills T, Seto TB, Sinclair KA. Cultural Dance Program Improves Hypertension Management for Native Hawaiians and Pacific Islanders: a Pilot Randomized Trial. J Racial Ethn Health Disparities. 2017 Feb;4(1):35-46. doi: 10.1007/s40615-015-0198-4. Epub 2015 Dec 22. PMID 27294768